CLINICAL TRIAL: NCT05552898
Title: Radicle™ Sleep: A Randomized, Blinded, Controlled, Direct-to-Consumer Study Assessing the Impact of Plant Derived Cannabinoids on Sleep and Overall Health Outcomes
Brief Title: Radicle Sleep: A Study of Plant Derived Cannabinoids on Sleep and Overall Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-22D01
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender and endorsement of problems with energy and/or focus reported during enrollment, then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo Control 1 (Placebo Comparator): Sleep Product Form 1 - control
  Interventions: Dietary Supplement: Sleep Study Product Usage
- Active Product 1.1 (Experimental): Sleep Product Form 1 - active product 1
  Interventions: Dietary Supplement: Sleep Study Product Usage
- Active Product 1.2 (Experimental): Sleep Product Form 1 - active product 2
  Interventions: Dietary Supplement: Sleep Study Product Usage
- Active Product 1.3 (Experimental): Sleep Product Form 1 - active product 3
  Interventions: Dietary Supplement: Sleep Study Product Usage
- Active Product 1.4 (Experimental): Sleep Product Form 1 - active product 4
  Interventions: Dietary Supplement: Sleep Study Product Usage
- Active Product 1.5 (Experimental): Sleep Product Form 1 - active product 5
  Interventions: Dietary Supplement: Sleep Study Product Usage

INTERVENTIONS:
Dietary Supplement: Sleep Study Product Usage — Participants will use their Radicle Sleep study product as directed for a period of 4 weeks.

SUMMARY:
A randomized, blinded, controlled, direct-to-consumer study assessing the impact of plant derived cannabinoids on sleep and overall health outcomes

DETAILED DESCRIPTION:
The aim of this study is to determine the safety and effects (if any) of different single agent and combination cannabinoid formulations on self-reported sleep and health in adults (21 years of age and older) that reside in the USA. It is a virtual, direct-to-consumer study that will recruit up to 300 participants per study arm (up to 1800 total). Participants will be followed for 5 weeks as they answer electronic surveys about their health, study product usage, and its impact on their health. There are no in-person visits for this study.

After study completion, study investigators will compare the effects of each cannabinoid study product to melatonin isolate. Study investigators will also run post-hoc analyses (correcting for multiple comparisons) to evaluate the significance of health score changes within individual study product arms, and whether there were significant differences in the effect with the addition of components to comparable cannabinoid study products.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Resides in the United States
* Endorses symptoms of sleep disturbance
* Selects sleep disturbance as a primary reason for taking a cannabinoid product
* Expresses a willingness to refrain from taking any non-study cannabinoid product (i.e. CBD, CBG, CBC, CBN, THC) for the duration of participant engagement (5 weeks)
* Expresses an interest in taking a study product and not knowing the product identity until the end of the study

Exclusion Criteria:

* Pregnant, trying to become pregnant, or breastfeeding
* Reports a diagnosis of liver disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Lack of reliable daily access to the internet
* Reports taking any medication that warns against grapefruit consumption

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1750 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Change in sleep disturbance | 4 weeks
  Sleep disturbance as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance SF 8A (Scoring from 8 to 40, with higher scores translating to greater sleep disturbance. Scores are standardized to US general population [T-score mapping])

SECONDARY OUTCOMES:
Change in sleep quantity | 4 weeks
  Sleep quantity as assessed by average hours of sleep reported per night
Change in overall well-being | 4 weeks
  Change in well-being as assessed by World Health Organization 5 (WHO-5 scale; Scoring from 0 to 25, with higher scores translating to greater well-being)
Change in anxiety | 4 weeks
  Anxiety as assessed by PROMIS Anxiety 4A (Scoring from 4 to 20, with higher scores translating to greater anxiety. Scores are standardized to US general population [T-score mapping)]
Change in pain | 4 weeks
  Pain as assessed by Pain on average, Enjoyment of life, and General activity Score (PEG; scale 0-10 where 0 is no pain)
Achievement of minimum clinically important difference (MCID) in sleep disturbance | 4 weeks
  Odds of achieving a MCID in sleep disturbance as assessed by Sleep disturbance as assessed by PROMIS Sleep Disturbance SF 8A

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com